CLINICAL TRIAL: NCT04578535
Title: A Phase 1, Open-Label, Randomized Study to Assess the Tolerability, Safety, and Pharmacokinetics of Subcutaneous Immune Globulin Infusion 10% (Human) With Recombinant Human Hyaluronidase (HYQVIA/HyQvia) With Ramp-Up and No Ramp-Up Dosing in Healthy Adult Subjects
Brief Title: A Study to Assess the Tolerability, Safety, and Pharmacokinetics of Subcutaneous Immune Globulin Infusion 10% (Human) With Recombinant Human Hyaluronidase (HYQVIA/HyQvia) With Ramp-up and No Ramp-up Dosing in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TAK-771-1001
Record Dates: First submitted 2020-07-07; First posted 2020-10-08 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1 Schedule A: TA 1 (Low TDL HYQVIA) (Experimental): Participants received a subcutaneous (SC) infusion of HYQVIA 0.1 g/kg (1/4 of TDL) on Day 1 and 8, 0.2 g/kg (1/2 of TDL) on Day 15, 0.3 g/kg (3/4 of TDL) on Day 29 followed by 0.4 g/kg (full TDL) on Day 50 in Ramp-Up dosing manner.
  Interventions: Drug: HYQVIA
- Part 2 Schedule A: TA 4 (High TDL HYQVIA) (Experimental): Participants received a SC infusion of HYQVIA 0.25 g/kg (1/4 of TDL) on Day 1 and 8, 0.5 g/kg (1/2 of TDL) on Day 15, 0.75 g/kg (3/4 of TDL) on Day 29 followed by 1.0 g/kg (full TDL) on Day 50 in Ramp-Up dosing manner.
  Interventions: Drug: HYQVIA
- Part 1 Schedule B: TA 2 (Low TDL HYQVIA) (Experimental): Participants received a SC infusion of HYQVIA 0.2 g/kg (1/2 of TDL) on Day 1 and 15, followed by 0.4 g/kg (full TDL) on Day 29 and 57 in Ramp-Up dosing manner.
  Interventions: Drug: HYQVIA
- Part 2 Schedule B: TA 5 (High TDL HYQVIA) (Experimental): Participants received a SC infusion of HYQVIA 0.5 g/kg (1/2 of TDL) on Day 1 and 15, followed by 1.0 g/kg (full TDL) on Day 29 and 57 in Ramp-Up dosing manner.
  Interventions: Drug: HYQVIA
- Part 1 Schedule C: TA 3 (Low TDL HYQVIA) (Experimental): Participants received a SC infusion of HYQVIA 0.4 g/kg (full TDL) SC infusion on Day 1, 29 and 57 without Ramp-Up dosing manner.
  Interventions: Drug: HYQVIA
- Part 2 Schedule C: TA 6 (High TDL HYQVIA) (Experimental): Participants received a SC infusion of HYQVIA 1.0 g/kg (full TDL) SC infusion on Day 1, 29 and 57 without Ramp-Up dosing manner.
  Interventions: Drug: HYQVIA

INTERVENTIONS:
Drug: HYQVIA — Participants received a SC infusion of HYQVIA 0.1 g/kg (1/4 of TDL) on Day 1 and 8, 0.2 g/kg (1/2 of TDL) on Day 15, 0.3 g/kg (3/4 of TDL) on Day 29 followed by 0.4 g/kg (full TDL) on Day 50 in Ramp-Up dosing manner.
  Other Names: IGI 10% with rHuPH20; Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase
  Arms: Part 1 Schedule A: TA 1 (Low TDL HYQVIA)
Drug: HYQVIA — Participants received a SC infusion of HYQVIA 0.25 g/kg (1/4 of TDL) on Day 1 and 8, 0.5 g/kg (1/2 of TDL) on Day 15, 0.75 g/kg (3/4 of TDL) on Day 29 followed by 1.0 g/kg (full TDL) on Day 50 in Ramp-Up dosing manner.
  Other Names: IGI 10% with rHuPH20; Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase
  Arms: Part 2 Schedule A: TA 4 (High TDL HYQVIA)
Drug: HYQVIA — Participants received a SC infusion of HYQVIA 0.2 g/kg (1/2 of TDL) on Day 1 and 15, followed by 0.4 g/kg (full TDL) on Day 29 and 57 in Ramp-Up dosing manner.
  Other Names: IGI 10% with rHuPH20; Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase
  Arms: Part 1 Schedule B: TA 2 (Low TDL HYQVIA)
Drug: HYQVIA — Participants received a SC infusion of HYQVIA 0.5 g/kg (1/2 of TDL) on Day 1 and 15, followed by 1.0 g/kg (full TDL) on Day 29 and 57 in Ramp-Up dosing manner.
  Other Names: IGI 10% with rHuPH20; Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase
  Arms: Part 2 Schedule B: TA 5 (High TDL HYQVIA)
Drug: HYQVIA — Participants received a SC infusion of HYQVIA 0.4 g/kg (full TDL) SC infusion on Day 1, 29 and 57 without Ramp-Up dosing manner.
  Other Names: IGI 10% with rHuPH20; Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase
  Arms: Part 1 Schedule C: TA 3 (Low TDL HYQVIA)
Drug: HYQVIA — Participants received a SC infusion of HYQVIA 1.0 g/kg (full TDL) SC infusion on Day 1, 29 and 57 without Ramp-Up dosing manner.
  Other Names: IGI 10% with rHuPH20; Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase
  Arms: Part 2 Schedule C: TA 6 (High TDL HYQVIA)

SUMMARY:
The purpose of the study is to assess the tolerability, safety, and pharmacokinetics of HYQVIA with ramp-up and no ramp-up dosing in healthy adult participants.

DETAILED DESCRIPTION:
This study will comprise of Part 1 and Part 2. Each study part will consist of three treatment arms (Part 1 [approximately 24 participants]: Treatment Arms 1-3 and Part 2 [approximately 24 participants]: Treatment Arms 4-6). Treatment arms will be initiated in parallel within each study part. Each participant will participate in only one treatment arm. After participants in Treatment Arms 1-3 (Study Part 1) will complete Week 9, the tolerability and, safety data through Week 9 will be reviewed by a safety review team. (Participants in arms 1-3 will continue in the study as the safety review is being completed.) Once the safety review for Arms 1-3 (Study part 1) will be completed and approved, Treatment Arms 4-6 (Study Part 2) will begin.

ELIGIBILITY:
Inclusion Criteria:

* An understanding, ability, and willingness to fully comply with study procedures and restrictions
* Ability to voluntarily provide written, signed, and dated (personally or via a legally authorized representative) informed consent to participate in the study
* Age 19-50 years inclusive at the time of consent. The date of signature of the informed consent is defined as the beginning of the screening period. This inclusion criterion will only be assessed at the first screening visit
* Male, or non-pregnant, non-breastfeeding female who agrees to comply with any applicable contraceptive requirements of the protocol, or females of non-childbearing potential
* Must be considered "healthy". Healthy as determined by the investigator on the basis of screening evaluations and healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electro cardiogram (ECG), hematology, blood chemistry, and urinalysis
* Body mass index (BMI) between 18.0 and 30.0 kilogram per square meter (kg/m^2) inclusive

Exclusion Criteria:

* Any current or relevant history of medical (e.g. any hematological, hepatic, respiratory, cardiovascular, renal or neurological) or psychiatric conditions, which by judgment of the investigator might compromise the safety of the participant or integrity of the study, interfere with the participant's participations in the trial and compromise the trial objectives or any condition that presents undue risk from the investigational product or procedures Note: Participants on stable dose of hormone replacements (i.e. thyroid hormone replacement) or oral contraceptives are permitted
* Clinically significant cardiac conditions including but not limited to uncontrolled hypertension, myocardial infarction, unstable coronary artery disease and clinically significant arrhythmias and conduction disorders
* Known or suspected intolerance or hypersensitivity to the investigational product(s), closely related compounds, or any of the stated ingredients (e.g. human IG, hyaluronidase, albumin)
* Known history of hypersensitivity or severe allergic reactions (e.g. urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following administration of blood or blood components
* Significant illness, as judged by the investigator, within 30 days of the first dose of investigational product
* Known history of alcohol or other substance abuse within the last year
* Donation of blood within 60 days, or blood products (e.g., plasma or platelets) within 2 weeks prior receiving the first dose of investigational product
* Participants will be excluded if any of the following laboratory parameters meet the criteria below:
* Hemoglobin less than (<) 11 gram per deciliter (g/dL). Absolute neutrophil count less than or equal to (< or =) 1500/ cubic millimeter (mm^3) and platelet count less than or equal to (< or =) 100,000/mm^3 Liver function: alanine aminotransferase (ALT) greater than or equal to > or =2.5 × upper limit normal (ULN), aspartate aminotransferase (AST) > or =2.5 × upper limit normal (ULN), alkaline phosphatase > or =1.5 × ULN or total bilirubin > or =1.5 milligram per deciliter (mg/dL) Renal function: creatinine clearance <or= 60 milliliter per minute (mL/min) based on Cockcroft-Gault equation Coagulation tests: activated partial thromboplastin time (aPTT) >1.2 X ULN; international normalized ratio (INR) >1.2 Participants will be excluded if any other laboratory values are outside the reference range and are clinically significant per investigator's judgment.
* Within 30 days prior to the first dose of investigational product:

  * Has participated in another clinical study involving immunoglobulin products within 12 months of screening.
  * Have used an investigational product (or 5 half-lives, whichever is longer).
  * Have been enrolled in a clinical study (including vaccine studies or has been vaccinated with approved product) that, in the investigator's opinion, may impact this study. Participants who have received any vaccine (including live attenuated vaccines) during the last 30 days before dosing will be excluded. No live attenuated virus vaccines are allowed during the study until the end of the follow up period
  * Have had any substantial changes in eating habits, as assessed by the investigator.
* Confirmed systolic blood pressure >139 mmHg or <89 mmHg and diastolic blood pressure >89 mmHg or <49 millimeters of Mercury (mmHg)
* A positive screen for alcohol or drugs of abuse at screening or D-1
* A positive human immunodeficiency virus (HIV), hepatitis C virus (HCV), or ongoing/active hepatitis B infection at screening. Participants with immunity to hepatitis B from either active vaccination or from previous natural infection are eligible to participate in the study.
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during confinement in the CRU
* Severe dermatitis or anatomical abnormality that would interfere with HYQVIA administration or endpoint assessments Note: the skin at the administration site should not be covered by tattoos.
* Current use of any herbal, or homeopathic preparations are not permitted
* Unable or unwilling to discontinue antihistamines or medications with antihistamine properties, sedatives, anxiolytics, systemic steroids, or topical steroids or antibiotics on any area below the chest for a minimum of 48 hours prior to each infusion visit and through 72 hours post last infusion
* Current or relevant history of hypercoagulable conditions (e.g. Protein C, Protein S, and antithrombin III deficiency), thrombotic/thromboembolic events or venous thrombosis

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- Clinical Pharmacology of Miami, Inc, Hialeah, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5facd1de17465c002989a195

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 participants were enrolled in the study, 33 participants into the Ramp-Up dosing group (treatment arms [TA] 1, 2, 4, and 5) and 18 participants into the No Ramp-Up dosing group (TA 3 and TA 6).
Pre-assignment Details: This study was conducted in 2 parts with a target dose level (TDL) of either 0.4 grams/kilograms (g/kg) (Part 1) or 1.0 g/kg (Part 2) through dose Ramp-Up or No Ramp-Up (direct administration of TDL). Each study part consisted of 3 TA (Part 1: TA 1 to 3 and Part 2: TA 4 to 6. TA 1 and 4 followed Schedule A (1/4 of the TDL to the full TDL) and TA 2 and 5 followed Schedule B (1/2 of TDL to full TDL) and TA 3 and 6 followed no ramp up (Schedule C).
Period: Overall Study
Arm/Group | Part 1 Schedule A: TA 1 (Low TDL HYQVIA) | Part 2 Schedule A: TA 4 (High TDL HYQVIA) | Part 1 Schedule B: TA 2 (Low TDL HYQVIA) | Part 2 Schedule B: TA 5 (High TDL HYQVIA) | Part 1 Schedule C: TA 3 (Low TDL HYQVIA) | Part 2 Schedule C: TA 6 (High TDL HYQVIA)
Started | 8 | 8 | 8 | 9 | 8 | 10
Completed | 6 | 8 | 8 | 7 | 6 | 3
Not Completed | 2 | 0 | 0 | 2 | 2 | 7
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 2
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 5
Not completed — Non-Compliance with Study Procedures | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all enrolled participants who received at least 1 dose of HYQVIA.
Groups:
- Part 1 Schedule A: TA 1 (Low TDL HYQVIA): Participants received a SC infusion of HYQVIA 0.1 g/kg (1/4 of TDL) on Day 1 and 8, 0.2 g/kg (1/2 of TDL) on Day 15, 0.3 g/kg (3/4 of TDL) on Day 29 followed by 0.4 g/kg (full TDL) on Day 50 in Ramp-Up dosing manner.
- Total: Total of all reporting groups
Arm/Group | Part 1 Schedule A: TA 1 (Low TDL HYQVIA) | Part 2 Schedule A: TA 4 (High TDL HYQVIA) | Part 1 Schedule B: TA 2 (Low TDL HYQVIA) | Part 2 Schedule B: TA 5 (High TDL HYQVIA) | Part 1 Schedule C: TA 3 (Low TDL HYQVIA) | Part 2 Schedule C: TA 6 (High TDL HYQVIA) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8 | 10 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (8.04) | 34.4 (6.44) | 40.4 (5.01) | 36.4 (7.88) | 36.8 (8.58) | 34.0 (10.07) | 35.1 (8.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 4 | 5 | 4 | 4 | 29
  Male | 1 | 3 | 4 | 4 | 4 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 6 | 9 | 6 | 10 | 47
  Not Hispanic or Latino | 0 | 0 | 2 | 0 | 2 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 4 | 3 | 2 | 2 | 17
  White | 4 | 6 | 4 | 6 | 6 | 8 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Tolerated All Initiated HYQVIA Infusion
Description: A tolerability event was considered to have occurred if an infusion was tolerable. An infusion was considered tolerable if the infusion rate was not reduced, or the infusion was not interrupted or stopped, due to an adverse event (AE) related to HYQVIA infusion. Tolerability was measured in terms of the number of participants for which the infusions was tolerable. Number of participants who tolerated all initiated HYQVIA Infusion were reported.
Time Frame: From start of the study drug administration up to Week 9
Population: The safety set included all enrolled participants who received at least 1 dose of HYQVIA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Schedule A: TA 1 (Low TDL HYQVIA) | Part 2 Schedule A: TA 4 (High TDL HYQVIA) | Part 1 Schedule B: TA 2 (Low TDL HYQVIA) | Part 2 Schedule B: TA 5 (High TDL HYQVIA) | Part 1 Schedule C: TA 3 (Low TDL HYQVIA) | Part 2 Schedule C: TA 6 (High TDL HYQVIA)
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8 | 10
Participants | 7 | 8 | 8 | 9 | 8 | 10

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events (TEAE) were defined as any event not present prior to the initiation of the treatments or any event already present that worsened in either intensity or frequency following exposure to the treatments. Number of participants with TEAEs was reported.
Time Frame: From start of the study drug administration up to Week 25
Population: The safety set included all enrolled participants who received at least 1 dose of HYQVIA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Schedule A: TA 1 (Low TDL HYQVIA) | Part 2 Schedule A: TA 4 (High TDL HYQVIA) | Part 1 Schedule B: TA 2 (Low TDL HYQVIA) | Part 2 Schedule B: TA 5 (High TDL HYQVIA) | Part 1 Schedule C: TA 3 (Low TDL HYQVIA) | Part 2 Schedule C: TA 6 (High TDL HYQVIA)
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8 | 10
Participants | 8 | 8 | 8 | 9 | 8 | 10

3. Secondary Outcome: Number of Participants Who Developed Binding and Neutralizing Antibodies to Recombinant Human Hyaluronidase PH20 (rHuPH20)
Description: Binding antibodies are responsible for binding to a pathogen and alerting the immune system to its presence so white blood cells can be sent to destroy it. The antibody level (titer) in the blood tells health care provider whether or not participant been exposed to an antigen, or something that the body thinks is foreign. A neutralizing antibody (NAb) is an antibody that is responsible for defending cells from pathogens, which are organisms that cause disease. The number of participants who developed binding and neutralizing antibodies to rHuPH20 were reported.
Time Frame: From start of the study drug administration up to Week 25
Population: The safety set included all enrolled participants who received at least 1 dose of HYQVIA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Schedule A: TA 1 (Low TDL HYQVIA) | Part 2 Schedule A: TA 4 (High TDL HYQVIA) | Part 1 Schedule B: TA 2 (Low TDL HYQVIA) | Part 2 Schedule B: TA 5 (High TDL HYQVIA) | Part 1 Schedule C: TA 3 (Low TDL HYQVIA) | Part 2 Schedule C: TA 6 (High TDL HYQVIA)
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8 | 10
Participants
  Binding ADA (Anti-Drug Antibodies) | 2 | 3 | 2 | 1 | 1 | 2
  Neutralizing ADA | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Time of Maximum Observed Serum Concentration (Tmax) of Total IgG and IgG Subclasses (IgG1, IgG2, IgG3, IgG4)
Description: Tmax was a measure of the time to reach the maximum concentration in the plasma after the drug dose. Summarized baseline corrected data was reported.
Time Frame: Pre-dose (Day 1), and 48, 96, 144 and 192 hours post-dose for all treatment arms; 360 hours post-dose for treatment arms 2 and 5; 360 and 696 hours post-dose for treatment arms 3 and 6
Population: PK Set included all enrolled participants received at least 1 dose of HYQVIA and had at least 1 evaluable post-dose serum concentration for total IgG or IgG subclasses. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable at the specified categories.
Measure: Median (Full Range); unit: days
Arm/Group | Part 1 Schedule A: TA 1 (Low TDL HYQVIA) | Part 2 Schedule A: TA 4 (High TDL HYQVIA) | Part 1 Schedule B: TA 2 (Low TDL HYQVIA) | Part 2 Schedule B: TA 5 (High TDL HYQVIA) | Part 1 Schedule C: TA 3 (Low TDL HYQVIA) | Part 2 Schedule C: TA 6 (High TDL HYQVIA)
Number analyzed (Participants) | 5 | 8 | 8 | 9 | 9 | 10
days
  Total IgG: number analyzed (Participants) | 2 | 5 | 3 | 9 | 7 | 10
  Total IgG | 5.0 [2.0 to 8.0] | 4.0 [2.0 to 8.0] | 8.0 [6.0 to 16.0] | 6.0 [4.0 to 16.1] | 4.0 [4.0 to 15.0] | 6.0 [4.0 to 8.0]
  Baseline corrected IgG1: number analyzed (Participants) | 2 | 6 | 8 | 8 | 9 | 10
  Baseline corrected IgG1 | 5.0 [4.0 to 6.0] | 5.0 [4.0 to 8.0] | 7.0 [4.0 to 15.0] | 7.0 [6.0 to 8.0] | 6.0 [6.0 to 8.0] | 6.0 [4.0 to 8.0]
  Baseline corrected IgG2: number analyzed (Participants) | 5 | 8 | 8 | 7 | 8 | 10
  Baseline corrected IgG2 | 6.0 [2.0 to 8.0] | 7.0 [2.0 to 8.0] | 8.0 [4.0 to 15.0] | 6.0 [4.0 to 8.0] | 7.0 [4.0 to 16.1] | 7.0 [4.0 to 15.0]
  Baseline corrected IgG3: number analyzed (Participants) | 2 | 3 | 6 | 3 | 8 | 10
  Baseline corrected IgG3 | 5.0 [4.0 to 6.0] | 8.0 [6.0 to 16.0] | 8.0 [4.0 to 15.0] | 4.0 [4.0 to 8.0] | 7.0 [2.0 to 16.1] | 5.0 [4.0 to 8.0]
  Baseline corrected IgG4: number analyzed (Participants) | 1 | 4 | 7 | 5 | 8 | 9
  Baseline corrected IgG4 | 4.0 [4.0 to 4.0] | 8.0 [2.0 to 8.0] | 8.0 [4.0 to 15.0] | 8.0 [4.0 to 8.0] | 7.0 [4.0 to 8.0] | 6.0 [4.0 to 8.0]

5. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) Sampled During a Dosing Interval of Total IgG and IgG Subclasses (IgG1, IgG2, IgG3, IgG4)
Description: Cmax was a measure of the maximum amount of drug in the serum after the dose is given. Summarized baseline corrected data was reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: grams per liter (g/L)
Arm/Group | Part 1 Schedule A: TA 1 (Low TDL HYQVIA) | Part 2 Schedule A: TA 4 (High TDL HYQVIA) | Part 1 Schedule B: TA 2 (Low TDL HYQVIA) | Part 2 Schedule B: TA 5 (High TDL HYQVIA) | Part 1 Schedule C: TA 3 (Low TDL HYQVIA) | Part 2 Schedule C: TA 6 (High TDL HYQVIA)
Number analyzed (Participants) | 5 | 8 | 8 | 9 | 9 | 10
grams per liter (g/L)
  Total IgG: number analyzed (Participants) | 2 | 5 | 3 | 9 | 7 | 10
  Total IgG | 2.70 (116.8) | 3.17 (66.8) | 3.10 (37.1) | 5.71 (41.0) | 5.34 (51.9) | 12.75 (16.2)
  Baseline corrected IgG1: number analyzed (Participants) | 2 | 6 | 8 | 8 | 9 | 10
  Baseline corrected IgG1 | 0.38 (58.5) | 1.51 (43.6) | 2.08 (25.1) | 1.11 (57.5) | 2.96 (36.2) | 5.88 (16.7)
  Baseline corrected IgG2: number analyzed (Participants) | 5 | 8 | 8 | 7 | 8 | 10
  Baseline corrected IgG2 | 0.48 (52.8) | 0.96 (52.6) | 1.33 (19.6) | 1.18 (74.8) | 1.98 (48.8) | 3.99 (41.9)
  Baseline corrected IgG3: number analyzed (Participants) | 2 | 3 | 6 | 3 | 8 | 10
  Baseline corrected IgG3 | 0.07 (5.7) | 0.03 (101.9) | 0.07 (26.4) | 0.04 (38.7) | 0.10 (67.6) | 0.19 (20.5)
  Baseline corrected IgG4: number analyzed (Participants) | 1 | 4 | 7 | 5 | 8 | 9
  Baseline corrected IgG4 | 0.02 | 0.08 (19.0) | 0.12 (46.8) | 0.13 (182.8) | 0.18 (32.7) | 0.29 (25.5)

6. Secondary Outcome: Area Under the Curve From the Time of Dosing to the Last Time Point With Measurable Concentration (AUClast) of Total IgG and IgG Subclasses (IgG1, IgG2, IgG3, IgG4)
Description: AUClast was a measure of the total amount of drug in the plasma from time zero to time of the last measurable concentration. Summarized baseline corrected data was reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*gram per liter (day*g/L)
Groups:
- Part 1 Schedule A: TA 1 (Low TDL HYQVIA): Participants received SC infusion of HYQVIA 0.1 g/kg (1/4 of TDL) on Day 1 and 8, 0.2 g/kg (1/2 of TDL) on Day 15, 0.3 g/kg (3/4 of TDL) on Day 29 followed by 0.4 g/kg (full TDL) on Day 50 in Ramp-Up dosing manner.
Arm/Group | Part 1 Schedule A: TA 1 (Low TDL HYQVIA) | Part 2 Schedule A: TA 4 (High TDL HYQVIA) | Part 1 Schedule B: TA 2 (Low TDL HYQVIA) | Part 2 Schedule B: TA 5 (High TDL HYQVIA) | Part 1 Schedule C: TA 3 (Low TDL HYQVIA) | Part 2 Schedule C: TA 6 (High TDL HYQVIA)
Number analyzed (Participants) | 5 | 8 | 8 | 9 | 8 | 10
day*gram per liter (day*g/L)
  Total IgG: number analyzed (Participants) | 2 | 5 | 3 | 9 | 7 | 10
  Total IgG | 9.63 (411.1) | 9.49 (39.0) | 31.60 (16.1) | 42.48 (43.3) | 70.39 (87.9) | 117.69 (65.5)
  Baseline corrected IgG1: number analyzed (Participants) | 2 | 6 | 8 | 8 | 8 | 10
  Baseline corrected IgG1 | 1.29 (46.6) | 11.37 (94.9) | 20.71 (60.1) | 4.30 (59.5) | 25.36 (51.6) | 60.04 (60.6)
  Baseline corrected IgG2: number analyzed (Participants) | 5 | 8 | 8 | 7 | 8 | 10
  Baseline corrected IgG2 | 1.66 (42.5) | 6.59 (102.1) | 17.36 (43.9) | 4.37 (49.7) | 17.77 (75.4) | 42.27 (86.3)
  Baseline corrected IgG3: number analyzed (Participants) | 2 | 3 | 6 | 3 | 8 | 10
  Baseline corrected IgG3 | 0.27 (27.4) | 0.22 (31.3) | 0.54 (79.0) | 0.17 (55.5) | 0.62 (90.5) | 1.33 (49.7)
  Baseline corrected IgG4: number analyzed (Participants) | 1 | 4 | 7 | 5 | 8 | 9
  Baseline corrected IgG4 | 0.06 | 0.40 (50.6) | 1.04 (45.8) | 0.39 (119.7) | 1.27 (75.3) | 2.43 (61.3)

7. Secondary Outcome: Terminal Half-Life (T1/2) of Total IgG and IgG Subclasses (IgG1, IgG2, IgG3, IgG4)
Description: T1/2 was the time required for a given drug concentration in the plasma to decrease by 50%. Summarized baseline corrected data was reported.
Time Frame: as for outcome 4
Population: PK Set included all enrolled participants received at least 1 dose of HYQVIA and had at least 1 evaluable post-dose serum concentration for total IgG or IgG subclasses. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable at the specified categories. "0" in analyzed field signifies that none of the participants had evaluable data at specified timepoint.
Measure: Median (Full Range); unit: days
Arm/Group | Part 1 Schedule A: TA 1 (Low TDL HYQVIA) | Part 2 Schedule A: TA 4 (High TDL HYQVIA) | Part 1 Schedule B: TA 2 (Low TDL HYQVIA) | Part 2 Schedule B: TA 5 (High TDL HYQVIA) | Part 1 Schedule C: TA 3 (Low TDL HYQVIA) | Part 2 Schedule C: TA 6 (High TDL HYQVIA)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0
days
  Total IgG |  |  |  |  | 8.1 [5.9 to 10.3] |
  Baseline corrected IgG1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Baseline corrected IgG2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Baseline corrected IgG3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Baseline corrected IgG4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Apparent Total Clearance After Extravascular Administration (CL/F) of Total IgG and IgG Subclasses (IgG1, IgG2, IgG3, IgG4)
Description: Apparent clearance was a calculation of the rate at which a drug is removed from plasma after oral administration via renal, hepatic and other clearance pathways, expressed as volume (milliliters) per unit of time (minutes). Summarized baseline corrected data was reported.
Time Frame: as for outcome 4
Population: PK Set included all enrolled participants received at least 1 dose of HYQVIA and had at least 1 evaluable post-dose serum concentration for total IgG or IgG subclasses. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "0" in analyzed field signifies that none of the participants had evaluable data at specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per day per kilograms (L/day/kg)
Groups:
- Part 2 Schedule B: TA 5 (High TDL HYQVIA): Participants received a SC infusion of HYQVIA 0.5 g/kg (1/2 of TDL) on days 1 and 15, followed by 1.0 g/kg (full TDL) at days 29 and 57 in Ramp-Up dosing manner.
Arm/Group | Part 1 Schedule A: TA 1 (Low TDL HYQVIA) | Part 2 Schedule A: TA 4 (High TDL HYQVIA) | Part 1 Schedule B: TA 2 (Low TDL HYQVIA) | Part 2 Schedule B: TA 5 (High TDL HYQVIA) | Part 1 Schedule C: TA 3 (Low TDL HYQVIA) | Part 2 Schedule C: TA 6 (High TDL HYQVIA)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0
liters per day per kilograms (L/day/kg)
  Total IgG |  |  |  |  | 0.01 (19.3) |
  Baseline corrected IgG1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Baseline corrected IgG2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Baseline corrected IgG3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Baseline corrected IgG4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Apparent Volume of Distribution Associated With the Terminal Slope Following Extravascular Administration (Vz/F) of Total IgG and IgG Subclasses (IgG1, IgG2, IgG3, IgG4)
Description: Volume of distribution (Vz/F) was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose is influenced by the fraction absorbed. Summarized baseline corrected data was reported.
Time Frame: as for outcome 4
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per kilogram (L/Kg)
Groups:
- Part 2 Schedule C: TA 6 (High TDL HYQVIA): Participants received a SC infusion of HYQVIA 1.0 g/kg (full TDL) SC infusion on Day 1, 29 and 57 without Ramp-Up dosing manner,
Arm/Group | Part 1 Schedule A: TA 1 (Low TDL HYQVIA) | Part 2 Schedule A: TA 4 (High TDL HYQVIA) | Part 1 Schedule B: TA 2 (Low TDL HYQVIA) | Part 2 Schedule B: TA 5 (High TDL HYQVIA) | Part 1 Schedule C: TA 3 (Low TDL HYQVIA) | Part 2 Schedule C: TA 6 (High TDL HYQVIA)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0
Liter per kilogram (L/Kg)
  Total IgG |  |  |  |  | 0.07 (20.6) |
  Baseline corrected IgG1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Baseline corrected IgG2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Baseline corrected IgG3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Baseline corrected IgG5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of the study drug administration up to Week 25
Description: The safety set included all enrolled participants who received at least 1 dose of HYQVIA.
Arm/Group | Part 1 Schedule A: TA 1 (Low TDL HYQVIA) | Part 2 Schedule A: TA 4 (High TDL HYQVIA) | Part 1 Schedule B: TA 2 (Low TDL HYQVIA) | Part 2 Schedule B: TA 5 (High TDL HYQVIA) | Part 1 Schedule C: TA 3 (Low TDL HYQVIA) | Part 2 Schedule C: TA 6 (High TDL HYQVIA)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/9 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/9 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8 | 9/9 | 8/8 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Schedule A: TA 1 (Low TDL HYQVIA) (N=8) | Part 2 Schedule A: TA 4 (High TDL HYQVIA) (N=8) | Part 1 Schedule B: TA 2 (Low TDL HYQVIA) (N=8) | Part 2 Schedule B: TA 5 (High TDL HYQVIA) (N=9) | Part 1 Schedule C: TA 3 (Low TDL HYQVIA) (N=8) | Part 2 Schedule C: TA 6 (High TDL HYQVIA) (N=10)
Blood pressure systolic decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 2 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2
Infusion site erythema (General disorders) | 5 | 6 | 5 | 9 | 6 | 10
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Infusion site pain (General disorders) | 3 | 5 | 6 | 9 | 5 | 7
Infusion site pruritus (General disorders) | 4 | 3 | 7 | 5 | 3 | 5
Infusion site swelling (General disorders) | 8 | 8 | 8 | 9 | 8 | 10
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT04578535/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT04578535/SAP_001.pdf